CLINICAL TRIAL: NCT06769165
Title: EMDR Treatment of Conditioned Nausea and Vomiting in Cancer Survivors - a Pilot Study
Brief Title: EMDR Treatment of Conditioned Nausea and Vomiting in Cancer Survivors
Acronym: EMESIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19946
Record Dates: First submitted 2024-12-09; First posted 2025-01-10 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Cancer Survivors
Keywords: EMDR; Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMDR Therapy (Experimental): EMDR therapy sessions with a trained psychologist.
  Interventions: Other: EMDR therapy

INTERVENTIONS:
Other: EMDR therapy — In this study, EMDR therapy will be performed by psychologists of the UMCG who are trained in EMDR therapy and who have experience with patients with somatic diseases. In the EMDR therapy protocol, the patient is guided through eight phases which incorporate dual focus of attention and alternating bilateral visual, auditory, and/or tactile stimulation (see supplement for protocol). The number of sessions varies per patient (1-3 sessions), depending on the desensitization of the conditioned stimuli. The sessions will last 60-90 minutes.

SUMMARY:
To explore the effectiveness of EMDR therapy treatment in reducing symptoms of chemotherapy-induced conditioned nausea and vomiting in (former) patients with cancer.

DETAILED DESCRIPTION:
Conditioned nausea and vomiting is a common side effect of anti-cancer treatment, and while strategies like antiemetics exist, their effectiveness is limited. Conditioned nausea and vomiting can possibly be addressed through Eye Movement Desensitization and Reprocessing (EMDR) therapy. EMDR therapy is a therapeutic intervention, proven to be effective in the treatment of post-traumatic stress disorder (PTSD), and promising in treating a range of other conditions. At the UMCG, EMDR therapy is used on a small scale to treat conditioned nausea with positive results, although more rigorous research is needed to fully establish its efficacy. This study aims to explore the effectiveness of EMDR therapy treatment in reducing symptoms of chemotherapy-induced conditioned nausea and vomiting in (former) patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Previously pathologically confirmed diagnosis of cancer
* Previously treated with systemic cancer therapy
* Persistent complaints (more than 2 months) of conditioned nausea and/or vomiting
* Able to understand spoken and written Dutch
* 18 years or older

Exclusion Criteria:

* Ongoing psychiatric treatment
* EMDR therapy contraindications (dissociative disorders, personality disorders or severe somatic disorders (e.g. cardiac arrhythmias))
* Complex type 2 trauma
* Known with recent conditions / non-anti-cancer medication which can elicit nausea (e.g. pregnancy or alcohol abuses)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Degree of conditioned nausea and vomiting | Before intake EMDR therapy session and three weeks after last EMDR therapy session
  Degree of conditioned nausea and vomiting after exposure to conditioned stimuli using the nausea profile questionnaire measured using the nausea profile questionnaire (9-point Likert scale, higher scores = worse outcome)

SECONDARY OUTCOMES:
Impact on QoL of conditioned nausea and vomiting | Before EMDR therapy
  Impact on QoL of conditioned nausea and vomiting using Functional Living Index- Emesis (FLIE) questionnaire (7-point Likert scale, higher scores = better/worse outcome, depending on the question)

CONTACTS AND LOCATIONS:
Overall Officials: Jacco J de Haan, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No